CLINICAL TRIAL: NCT05120947
Title: A Phase I Study of Hypofractionated Adjuvant Radiotherapy for Resected Head and Neck Cancers (HART-HN)
Brief Title: Hypofractionated Adjuvant Radiotherapy for Resected Head and Neck Cancers
Acronym: HART-HN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Musaddiq Awan, Assistant Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO00042119
Record Dates: First submitted 2021-11-03; First posted 2021-11-16 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Resectable Head and Neck Squamous Cell Carcinoma
Keywords: Head and Neck Squamous Cell Carcinoma; Hypofraction Adjuvant Radiation
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: This study will use a time-to-event continual reassessment method (TITE-CRM) for assigning subjects to the radiation therapy dosages.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- 42 Gray (Gy) Radiation (Experimental): 42 gy of radiation therapy will be administered in 10 fractions.
  Interventions: Radiation: 42 Gy Radiation Therapy
- 39 Gray (Gy) Radiation (Experimental): 39 gy of radiation therapy will be administered in 8 fractions.
  Interventions: Radiation: 39 Gy Radiation Therapy
- 32.5 Gray (Gy) Radiation (Experimental): 32.5 gy of radiation therapy will be administered in 5 fractions.
  Interventions: Radiation: 32.5 Gy Radiation Therapy

INTERVENTIONS:
Radiation: 42 Gy Radiation Therapy — Radiation Therapy: Dose per fraction of 4.2 Gy.
  Arms: 42 Gray (Gy) Radiation
Radiation: 39 Gy Radiation Therapy — Radiation Therapy: Dose per fraction of 4.875 Gy.
  Arms: 39 Gray (Gy) Radiation
Radiation: 32.5 Gy Radiation Therapy — Radiation Therapy: Dose per fraction of 6.5 Gy.
  Arms: 32.5 Gray (Gy) Radiation

SUMMARY:
The primary purpose of this study is to determine the safe reduction of the treatment fractions to 10, 8, or 5, that may be delivered safely in resected head and neck squamous cell carcinoma (HNSCC) patients with intermediate pathologic risk features.

DETAILED DESCRIPTION:
RATIONALE: Postoperative hypofractionated radiation is well established in many malignancies, yielding benefits in compliance, access to care, convenience, and cost savings. In several solid tumor types, short-course high dose-per-fraction (hypofractionated) post-operative radiation has shown excellent tolerability, reduced healthcare costs, improved compliance, and at least equivalent cancer control compared to conventional post-operative radiation (long course, low dose-per-fraction).(1-3) Despite advances in other malignancies, hypofractionated post-operative radiation is not used in previously untreated mucosal HNSCCs, for which an extended course of conventional post-operative radiation (usually 60 Gy in 2 Gy fractions delivered over six weeks) remains the standard. Hypofractionation has been stymied in the post-operative setting for HNSCCs primarily due to concerns of toxicity in treating a large mucosal field and an inability to spare critical structures such as the brain and spinal cord. These concerns were well-founded in the 1970s during the era of 2-dimensional radiotherapy when conventional HNSCC radiotherapy regimens were developed.(4) But because radiotherapy can be delivered far more precisely using intensity modulated radiation therapy (IMRT), it is hypothesized that post-operative radiation for HNSCCs can now be delivered safely in only five fractions delivered over one week.(3, 5, 6)

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older with gross totally resected (R0 resection) Human papillomavirus (HPV) -negative squamous cell carcinoma of the head and neck (squamous cell carcinoma of the larynx, hypopharynx, oropharynx, oral cavity, nasal cavity, paranasal sinuses or carcinoma of unknown head/neck primary) who have at least 1 of the following intermediate risk factors for adjuvant radiation:

   1. Pathologic Node Positive Disease
   2. Perineural Invasion
   3. Oral cavity cancer with depth of invasion of at least 5 mm
   4. Lymphovascular Space Invasion
   5. Pathologic T3 or T4 disease
2. Zubrod performance status 0-2.
3. Patients must have the psychological ability and general health that permits completion of the study requirements and required follow up.
4. Inclusion of Covid-19 positive patients will be based on standard institutional protocol.
5. Female patients must meet one of the following:

   * Postmenopausal for at least one year before the screening visit, or
   * Surgically sterile (i.e. undergone a hysterectomy or bilateral oophorectomy), or
   * If subject is of childbearing potential (defined as not satisfying either of the above two criteria), agree to practice two acceptable methods of contraception (combination methods requires use of two of the following: diaphragm with spermicide, cervical cap with spermicide, contraceptive sponge, male or female condom, hormonal contraceptive) from the time of signing of the informed consent form through 90 days after the last dose of study agent, AND o Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptom-thermal, post ovulation methods] and withdrawal are not acceptable contraception methods).
6. Male patients, even if surgically sterilized (i.e., status post vasectomy), must agree to one of the following:

   * Practice effective barrier contraception during the entire study period and through 60 calendar days after the last dose of study agent, OR
   * Must also adhere to the guidelines of any study-specific pregnancy prevention program, if applicable, OR o Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptom-thermal, post ovulation methods] and withdrawal are not acceptable methods of contraception.)
7. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Pathologic evidence of extranodal extension.
2. Pathologic evidence of a final positive margin (R1 resection) or gross residual disease (R2 resection).
3. HPV-positive squamous cell carcinoma.
4. Prior invasive malignancy within the past 3 years (except for non-melanomatous skin cancer, and early stage treated prostate cancer).
5. Life expectancy less than 12 months.
6. Performance status Zubrod ≥ 3.
7. Patients with prior radiation therapy to the head and neck Note: Prior external beam radiotherapy is excluded, but Iodine 131 is allowed.
8. Prior systemic therapy, including cytotoxic chemotherapy, biologic/targeted therapy, or immune therapy for the study cancer.
9. Body weight ≤ 30 kg.
10. Any of the following severe laboratory abnormalities within 14 days of registration, unless corrected prior to it: Sodium < 130 mmol/L or > 155 mmol/L; Potassium < 3.5 mmol/L or > 6 mmol/L; Fasting glucose < 40 mg/dl or > 400 mg/dl; Serum calcium (ionized or adjusted for albumin) < 7 mg/dl or > 12.5 mg/dl; Magnesium < 0.9 mg/dl or > 3 mg/dl.
11. Unstable angina and/or congestive heart failure requiring hospitalization within 3 months prior to Step 1 registration.
12. Transmural myocardial infarction within three months prior to Step 1 registration.
13. Medical or psychiatric illness which would compromise the patient's ability to tolerate treatment or limit compliance with study requirements.
14. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception during treatment and for 6 months after radiation, this exclusion is necessary because the treatment involved in this study may be significantly teratogenic. Women who are breastfeeding are also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-11-22 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated Radiation Dose | 12 months
  This will be determined as the radiation dose with the minimum number of fractions at which there is no more than a 33% rate of dose-limiting toxicity (DLT) up to 12 months after completion of radiation treatment using the TITE-CRM design.
Incidence of Dose-Limiting Toxicities | 12 months
  This measure is the number of subjects experiencing a dose-limiting toxicity. A dose-limiting toxicity is defined as an inability to complete radiation treatment within 30 days of the start of radiotherapy that is not deemed to be related to disease progression; OR an unacceptable toxicity within one year of treatment (Grade 4+ toxicity) that is probably or definitely related to radiation treatment as determined by the treating physician or a death within one year of treatment that is probably or definitely related to treatment.

SECONDARY OUTCOMES:
Overall Survival | One year
  This measure is the number of subjects alive at one year following the conclusion of scheduled radiation therapy.
Locoregional progression | One year
  This measure is the number of subjects showing disease progression in the head and neck by response evaluation criteria in solid tumors (RECIST) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Musaddiq Awan, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moran MS, Truong PT. Hypofractionated radiation treatment for breast cancer: The time is now. Breast J. 2020 Jan;26(1):47-54. doi: 10.1111/tbj.13724. Epub 2020 Jan 15. PMID 31944484
- [Background] Benjamin LC, Tree AC, Dearnaley DP. The Role of Hypofractionated Radiotherapy in Prostate Cancer. Curr Oncol Rep. 2017 Apr;19(4):30. doi: 10.1007/s11912-017-0584-7. PMID 28343352
- [Background] Stevens G, Thompson JF, Firth I, O'Brien CJ, McCarthy WH, Quinn MJ. Locally advanced melanoma: results of postoperative hypofractionated radiation therapy. Cancer. 2000 Jan 1;88(1):88-94. doi: 10.1002/(sici)1097-0142(20000101)88:13.0.co;2-k. PMID 10618610
- [Background] Tupchong L, Scott CB, Blitzer PH, Marcial VA, Lowry LD, Jacobs JR, Stetz J, Davis LW, Snow JB, Chandler R, et al. Randomized study of preoperative versus postoperative radiation therapy in advanced head and neck carcinoma: long-term follow-up of RTOG study 73-03. Int J Radiat Oncol Biol Phys. 1991 Jan;20(1):21-8. doi: 10.1016/0360-3016(91)90133-o. PMID 1993628
- [Background] Kumar AMS, Miller J, Hoffer SA, Mansur DB, Coffey M, Lo SS, Sloan AE, Machtay M. Postoperative hypofractionated stereotactic brain radiation (HSRT) for resected brain metastases: improved local control with higher BED10. J Neurooncol. 2018 Sep;139(2):449-454. doi: 10.1007/s11060-018-2885-6. Epub 2018 May 10. PMID 29749569
- [Background] Murray Brunt A, Haviland JS, Wheatley DA, Sydenham MA, Alhasso A, Bloomfield DJ, Chan C, Churn M, Cleator S, Coles CE, Goodman A, Harnett A, Hopwood P, Kirby AM, Kirwan CC, Morris C, Nabi Z, Sawyer E, Somaiah N, Stones L, Syndikus I, Bliss JM, Yarnold JR; FAST-Forward Trial Management Group. Hypofractionated breast radiotherapy for 1 week versus 3 weeks (FAST-Forward): 5-year efficacy and late normal tissue effects results from a multicentre, non-inferiority, randomised, phase 3 trial. Lancet. 2020 May 23;395(10237):1613-1626. doi: 10.1016/S0140-6736(20)30932-6. Epub 2020 Apr 28. PMID 32580883